CLINICAL TRIAL: NCT05737303
Title: Nab-paclitaxel Versus Solvent-based Taxanes As First-Line Treatment for Patients With Advanced Ovarian Cancer
Brief Title: Nab-paclitaxel Versus Sb-taxanes As First-Line Treatment in Advanced Ovarian Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Collaborators: Jiaxing Maternity and Child Health Care Hospital (Other); Zhejiang University (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Sun Yat-sen University (Other); Qilu Hospital of Shandong University (Other); Ningbo No. 1 Hospital (Other); Ningbo Women & Children's Hospital (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IRB-20230058-R
Record Dates: First submitted 2023-01-02; First posted 2023-02-21 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2024-11

CONDITIONS: Epithelial Ovarian Carcinoma Stage III; Epithelial Ovarian Carcinoma Stage IV; Fallopian Tube Carcinoma Stage III; Fallopian Tube Carcinoma Stage IV; Primary Peritoneal Carcinoma Stage III; Primary Peritoneal Carcinoma Stage IV
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Fallopian Tube Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nab-Paclitaxel/carboplatin for systemic therapy after surgery (Experimental): Nab-Paclitaxel/carboplatin q3 weeks Nab-Paclitaxel 260 mg/m² IV followed by carboplatin AUC（area under the curve） 5 IV Day1 Repeat every 21 days x 6 cycles Nab-Paclitaxel/carboplatin weekly Dose-dense Nab-Paclitaxel 100 mg/m2 IV followed by carboplatin AUC（area under the curve）2 IV Davs 1. 8, and 15 ·Repeat every 21 days x 6 cycles
  Interventions: Drug: nab-paclitaxel combined with carboplatin
- Paclitaxel/carboplatin for systemic therapy (Active Comparator): Paclitaxel 175 mg/m² IV followed by carboplatin AUC（area under the curve）5 IV Day·1Repeat every 21 days x 6 cycles
  Paclitaxel weekly/carboplatin weekly Paclitaxel 60 mg/m2 followed by carboplatin AUC（area under the curve） 2 IV Days 1.8. and 15: repeat every 21 days 6 cycles (18 weeks)
  Interventions: Drug: nab-paclitaxel combined with carboplatin

INTERVENTIONS:
Drug: nab-paclitaxel combined with carboplatin — Nab-Paclitaxel/carboplatin q3weeks Nab-Paclitaxel 260 mg/m² IV followed by carboplatin AUC（area under the curve） 5 IV Day1 Repeat every 21 days x 6 cycles Nab-Paclitaxel/carboplatin weekly Dose-dense Nab-Paclitaxel 100 mg/m2 IV followed by carboplatin AUC（area under the curve）2 IV Davs 1. 8, and 15 ·Repeat every 21 days x 6 cycles Paclitaxel 175 mg/m² IV followed by carboplatin AUC（area under the curve）5 IV Day·1Repeat every 21 days x 6 cycles
  Paclitaxel weekly/carboplatin weekly Paclitaxel 60 mg/m2 followed by carboplatin AUC（area under the curve）2 IV Days 1.8. and 15: repeat every 21 days 6 cycles (18 weeks)
  Other Names: paclitaxel combined with carboplatin

SUMMARY:
The purpose of this study is to compare the efficacy and safety of nab-paclitaxel with solvent-based taxanes as first-line treatment for patients with advanced primary epithelial ovarian cancer (EOC), primary peritoneal carcinoma or fallopian tube carcinoma.

DETAILED DESCRIPTION:
One of the major challenges related to solvent-based taxanes administration in clinical practice is the high rate of hypersensitivity reactions (HSRs). Nab-paclitaxel has showed its considerable survival and low toxicity profiles in first-line treatment for several solid tumors and is recommended as a treatment for recurrent epithelial ovarian cancer (EOC). We focus on clinical efficacy and safety outcomes of nab-paclitaxel in current clinical studies of primary EOC treatment and aim to explore the potential feasibility of nab-paclitaxel as the first-line treatment for EOC, primary peritoneal carcinoma or fallopian tube carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. Epithelial ovarian cancer/tubal cancer/peritoneal cancer was diagnosed by histopathology or hydroexfoliation cytopathology of the chest and abdomen, and was classified as stage III-IV according to FIGO（International Federation of Gynecology and Obstetrics）stage
2. Physical condition Eastern Cooperative Oncology Group PS score: 0-2 points
3. Participants who had not participated in other drug clinical trials within 4 weeks prior to enrollment
4. Written informed consent
5. Expected survival ≥6 months
6. The disease met the criteria for Efficacy Evaluation of solid tumors (RECIST 1.1)
7. Be able to comply with outpatient treatment, laboratory monitoring, and necessary clinical visits during study participation.

Exclusion Criteria:

1. Patients with low malignant potential ovarian tumors;
2. Other malignant tumors within the previous 5 years, except for cured cervical carcinoma in situ and non-melanoma skin cancer;
3. Patients who have previously received chemotherapy or radiotherapy for pelvic cavity;
4. Patients with central nervous system metastasis or peripheral neuropathy > grade 1;
5. Patients with severe myelosuppression, severe liver dysfunction (Child's Class III), or renal dysfunction at the time of screening;
6. Severe cardiovascular disease: Grade Ⅱ or above myocardial ischemia or myocardial infarction, poorly controlled arrhythmias (including QTc interval ≥470 ms); According to NYHA（New York Heart Association） criteria, patients with grade Ⅲ to Ⅳ cardiac insufficiency or left ventricular ejection fraction (LVEF) < 55% indicated by color Doppler ultrasonography;
7. Uncontrolled systemic infection requiring anti-infective treatment;
8. Arteriovenous thrombosis events occurring within 6 months before randomization, such as cardiovascular and cerebrovascular accidents (including temporary ischemic attack, cerebral hemorrhage, cerebral infarction, myocardial infarction), deep vein thrombosis and pulmonary embolism;
9. Patients who are allergic to the active ingredients or excipients of albumin paclitaxel and carboplatin for injection;
10. Pregnant or lactating women;
11. Those who were considered unsuitable for inclusion by the researchers.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 538 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 20 months
  Disease progression as first failure

SECONDARY OUTCOMES:
Objective Remission Rate | 12 months
  The target lesion disappeared for at least 4 weeks,Tumor volume reduced by at least 30 percent.
Survival | 3 years, 5 years
  Overall survival (all-cause death)
Adverse events | 3 years, 5 years
  Treatment-related symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Yaxia Chen, MD, Principal Investigator — Study Principal Investigator
Locations (11):
- China (11):
  - Sun Yat-Sen University Cancer Hospital, Guangzhou, Guangdong
  - Qilu Hospital of Shandong University, Ji'nan, Shandong
  - Yaxia Chen, Hangzhou, Zhejiang
  - Sir Run Run Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Medical College of Zhejiang University, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Ningbo women's and children's Hospital, Ningbo, Zhejiang
  - The No, 1 People's Hospital of Ningbo, Ningbo, Zhejiang
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Zheng L, Cui C, Shi O, Lu X, Li YK, Wang W, Li Y, Wang Q. Incidence and mortality of ovarian cancer at the global, regional, and national levels, 1990-2017. Gynecol Oncol. 2020 Oct;159(1):239-247. doi: 10.1016/j.ygyno.2020.07.008. Epub 2020 Jul 18. PMID 32690392
- [Background] Zeighami S, Soltani M, Khajeh F, Ariafar A, Naghdi-Sedeh N. Testicular papillary serous carcinoma of ovarian type, a rare case report, however an important timely diagnostic issue. Urol Case Rep. 2020 Jun 16;33:101301. doi: 10.1016/j.eucr.2020.101301. eCollection 2020 Nov. PMID 33102004
- [Background] Dueckelmann AM, Fink D, Harter P, Heinzelmann V, Marth C, Mueller M, Reinthaller A, Tamussino K, Wimberger P, Sehouli J. The use of PIPAC (pressurized intraperitoneal aerosol chemotherapy) in gynecological oncology: a statement by the "Arbeitsgemeinschaft Gynaekologische Onkologie Studiengruppe Ovarialkarzinom (AGO-OVAR)", the Swiss and Austrian AGO, and the North-Eastern German Society of Gynaecologic Oncology. Arch Gynecol Obstet. 2018 Apr;297(4):837-846. doi: 10.1007/s00404-018-4673-0. Epub 2018 Jan 22. PMID 29356953
- [Background] Perez-Fidalgo JA, Grau F, Farinas L, Oaknin A. Systemic treatment of newly diagnosed advanced epithelial ovarian cancer: From chemotherapy to precision medicine. Crit Rev Oncol Hematol. 2021 Feb;158:103209. doi: 10.1016/j.critrevonc.2020.103209. Epub 2020 Dec 31. PMID 33388455
- [Background] Huang CY, Cheng M, Lee NR, Huang HY, Lee WL, Chang WH, Wang PH. Comparing Paclitaxel-Carboplatin with Paclitaxel-Cisplatin as the Front-Line Chemotherapy for Patients with FIGO IIIC Serous-Type Tubo-Ovarian Cancer. Int J Environ Res Public Health. 2020 Mar 26;17(7):2213. doi: 10.3390/ijerph17072213. PMID 32224896
- [Background] Ozols RF, Bundy BN, Greer BE, Fowler JM, Clarke-Pearson D, Burger RA, Mannel RS, DeGeest K, Hartenbach EM, Baergen R; Gynecologic Oncology Group. Phase III trial of carboplatin and paclitaxel compared with cisplatin and paclitaxel in patients with optimally resected stage III ovarian cancer: a Gynecologic Oncology Group study. J Clin Oncol. 2003 Sep 1;21(17):3194-200. doi: 10.1200/JCO.2003.02.153. Epub 2003 Jul 14. PMID 12860964
- [Background] Ratanajarusiri T, Sriuranpong V, Sitthideatphaiboon P, Poovoravan N, Vinayanuwat C, Parinyanitikul N, Angspatt P, Thawinwisan W, Tanasanvimon S. A Difference in the Incidences of Hypersensitivity Reactions to Original and Generic Taxanes. Chemotherapy. 2017;62(2):134-139. doi: 10.1159/000450748. Epub 2016 Dec 20. PMID 27997900
- [Background] Kundranda MN, Niu J. Albumin-bound paclitaxel in solid tumors: clinical development and future directions. Drug Des Devel Ther. 2015 Jul 24;9:3767-77. doi: 10.2147/DDDT.S88023. eCollection 2015. PMID 26244011
- [Background] du Bois A, Quinn M, Thigpen T, Vermorken J, Avall-Lundqvist E, Bookman M, Bowtell D, Brady M, Casado A, Cervantes A, Eisenhauer E, Friedlaender M, Fujiwara K, Grenman S, Guastalla JP, Harper P, Hogberg T, Kaye S, Kitchener H, Kristensen G, Mannel R, Meier W, Miller B, Neijt JP, Oza A, Ozols R, Parmar M, Pecorelli S, Pfisterer J, Poveda A, Provencher D, Pujade-Lauraine E, Randall M, Rochon J, Rustin G, Sagae S, Stehman F, Stuart G, Trimble E, Vasey P, Vergote I, Verheijen R, Wagner U; Gynecologic Cancer Intergroup; AGO-OVAR; ANZGOG; EORTC; GEICO; GINECO; GOG; JGOG; MRC/NCRI; NCIC-CTG; NCI-US; NSGO; RTOG; SGCTG; IGCS; Organizational team of the two prior International OCCC. 2004 consensus statements on the management of ovarian cancer: final document of the 3rd International Gynecologic Cancer Intergroup Ovarian Cancer Consensus Conference (GCIG OCCC 2004). Ann Oncol. 2005;16 Suppl 8:viii7-viii12. doi: 10.1093/annonc/mdi961. No abstract available. PMID 16239238
- [Background] Wang H, Fan L, Wu X, Han Y. Efficacy evaluation of albumin-bound paclitaxel combined with carboplatin as neoadjuvant chemotherapy for primary epithelial ovarian cancer. BMC Womens Health. 2022 Jun 11;22(1):224. doi: 10.1186/s12905-022-01794-y. PMID 35690772
- [Background] Teneriello MG, Tseng PC, Crozier M, Encarnacion C, Hancock K, Messing MJ, Boehm KA, Williams A, Asmar L. Phase II evaluation of nanoparticle albumin-bound paclitaxel in platinum-sensitive patients with recurrent ovarian, peritoneal, or fallopian tube cancer. J Clin Oncol. 2009 Mar 20;27(9):1426-31. doi: 10.1200/JCO.2008.18.9548. Epub 2009 Feb 17. PMID 19224848